CLINICAL TRIAL: NCT04247165
Title: LAPTOP: Phase 1/2 Study in Borderline Resectable, Locally Advanced or Metastatic Pancreatic Cancer to Assess Safety and Potential Efficacy of Dual Checkpoint Inhibition in Combination with Gemcitabine and Nab-paclitaxel Followed by Immune-chemoradiation.
Brief Title: Nivolumab, Ipilimumab and Chemoradiation in Pancreatic Cancer.
Acronym: LAPTOP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Inna Chen, MD, Principal investigator, Herlev Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI 1931
Record Dates: First submitted 2020-01-25; First posted 2020-01-29 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-05

CONDITIONS: Borderline Resectable, Locally Advanced or Metastatic Pancreatic Cancer
Keywords: pancreatic cancer; borderline resectable, locally advanced or metastatic pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Nivolumab 3 mg/kg will be given on day 1 (± 2 days) of each 28-day treatment cycle until the progression of disease, discontinuation due to toxicity, withdrawal of consent. Ipilimumab 1 mg/kg will be given once only on day 1 cycle 1. Nivolumab will be administered as an IV infusion over 30 (± 5) minutes and then, after a 30 minutes rest period, ipilimumab will be administered as an IV infusion over 30 (± 5) minutes. Pre-medication for chemotherapy (based on standard-of-care and local institutional standards) and chemotherapy will then be administered after a further 30 minutes rest period.
  The recommended dose of nab-paclitaxel is 100 mg/m2 administered as an IV infusion over 30 to 40 minutes on Days 1, 8, and 15 of each 28-day cycle. Gemcitabine 800 mg/m2 will be administered over 30 to 40 minutes immediately after nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Nivolumab; Drug: Ipilimumab; Radiation: SBRT

INTERVENTIONS:
Drug: Gemcitabine — 800 mg/m2 Day 1, 8, 15: Q4W IV Infusion
Drug: Nab-paclitaxel — 100 mg/m2 Day 1, 8, 15: Q4W IV Infusion
  Other Names: Abraxane®
Drug: Nivolumab — 3 mg/kg Day 1, Q4W IV Infusion
  Other Names: Opdivo®
Drug: Ipilimumab — 1 mg/kg Day 1 Cycle 1 IV Infusion
  Other Names: Yervoy®
Radiation: SBRT — Patients will be planned and treated with SBRT on a MRidian MR guided Linac.
  Prescription dose shall be according to the following specifications:
  * Prescription dose shall be according to the following specifications:
  * A total dose of 24 Gy in 3 fractions (3 fractions/week) are prescribed as the mean dose to the PTV.
  * Pauses are accepted but the treatment should be delivered within 10 calendar days.
  * PTV should be covered by 95% isodose (PTV D99% >95%).

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) remains a dreadful disease due to its often advanced stage at diagnosis and poor sensitivity to chemotherapy. A locally unresectable tumor (locally advanced pancreatic cancer (LAPC)) is present in 30% of the cases and is defined as a surgically unresectable tumor encasing the adjacent arteries [celiac axis, superior mesenteric artery (SMA)]. In these patients, chemotherapy has been the standard treatment for decades, optionally combined with radiotherapy. Patients with borderline resectable pancreatic cancer (BRPC) comprise a group of patients with PDAC who are at a high risk of having positive margins if upfront resection is pursued. In addition, multiple studies have reported these patients have increased probability of early recurrence of local and systemic disease resulting in poorer outcomes. Although some patients are treated with an aggressive surgery-first approach and adjuvant systemic therapies, a preoperative chemotherapy and/or chemoradiation approach is becoming more common for all patients with BRPC, and this strategy is adapted in Danish and international guidelines. Majority of patients present with metastatic pancreatic cancer (mPC). Therapy options are limited by chemotherapy in palliative setting. The superiority of the FOLFIRINOX regimen demonstrated in the phase III mPC setting led many centers to investigate FOLFIRINOX with or without chemoradiotherapy in patients with LAPC tumor. Gemcitabine combined with nab-paclitaxel is the approved first-line treatment for patients with advanced PC. This regimen showed a median progression-free survival (PFS) of 5.5 months and a median overall survival (OS) of 8.5 months and is the predominantly used regimen in metastatic PC. The role of radiation therapy in the management of nonresectable PC remains controversial. The results of small randomized trials comparing chemoradiotherapy with chemotherapy of patients with LAPC are divergent.

Immunotherapy has emerged as a therapeutic approach that offers effective and durable treatment options for subsets of patients with various types of cancer. However, these successes have not manifested similar benefits for PDAC patients mostly due to a lack of pre-existing T-cell immunity and/or a highly immunosuppressive tumor microenvironment (TME). Considering the emerging role of the TME, the combination of checkpoint blocking antibodies with agents that target the inhibitory effects of the TME could lead to better responses in tumor historically resistant to checkpoint blocking antibody approaches. For example, in heavily pretreated patients with advanced/metastatic PDAC, preliminary data from the phase 2 study CHECKPAC (NCT02866383) showed that checkpoint inhibition in combination with stereotactic body radiotherapy (SBRT) provided durable clinical benefit in a small proportion of patients, including prolonged, sustained partial responses. Furthermore, the addition of standard-of-care chemotherapy could further potentiate the anti-tumor effects of immunotherapy approaches by reducing the tumor burden, exposing antigens, and directly affecting the immunosuppressive TME compartment.

To explore the safety and synergy of the proposed combinatorial approach, participants with borderline resectable, locally advanced or mPC will receive nivolumab and ipilimumab administered in combination with gemcitabine and nab-paclitaxel followed by immune-chemoradiation.

DETAILED DESCRIPTION:
Patients receive nivolumab and ipilimumab. Nivolumab 3 mg/kg will be given on Day 1 (± 3 days) of each 28-day treatment cycle. Ipilimumab 1 mg/kg will be given only on day 1 in cycle 1. Nivolumab will be administered as an IV infusion over 30 (± 5) minutes and then, after a 30 minutes rest period, ipilimumab will be administered as an IV infusion over 30 (± 5) minutes.

Pre-medication for chemotherapy (based on standard-of-care and local institutional standards) and chemotherapy will then be administered after a further 30 minutes rest period. The recommended dose of nab-paclitaxel is 100 mg/m2 administered as an IV infusion over 30 to 40 minutes on Days 1, 8, and 15 of each 28-day cycle. Gemcitabine 800 mg/m2 will be adminestered over 30 to 40 minutes immediately after nab-paclitaxel on Days 1, 8, and 15 of each 28-day cycle.

At the beginning of cycle 3, patients also undergo concurrent MRI-guided adaptive SBRT (8 Gy x 3 fractions) delivered by ViewRay MR-Linear Accelerator.

Cycles repeats every 4 weeks for 4 courses (16 weeks) in the absence of disease progression, unacceptable toxicity, withdrawal of consent, or study closure.

Once 4 cycles of study treatment have been completed, subjects without disease progression or unacceptable toxicity may continue as per Investigator's Choice to either:

* Continuation of treatment with nivolumab, nab-paclitaxel and gemcitabine or surgery. Nivolumab can be continued until progressive disease (PD), unacceptable toxicity, withdrawal of consent, or up to 12 cycles in total. Patients will receive chemotherapy until PD, unacceptable toxicity or withdrawal of consent, according to investigator's judgment
* If tumor response allows for surgical intervention, the subject will be eligible for that treatment as deemed appropriate by the investigators. Surgical intervention may not occur prior to completing the planned 4 cycles of nivolumab, nab-paclitaxel, gemcitabine and SBRT regardless the patient demonstrates a major response to therapy. Patients after PC resection will receive treatment until recurrence, unacceptable toxicity, withdrawal of consent, clear clinical deterioration, or for a maximum of 6 cycles, according to investigator's judgment Patients who discontinue without PD (stable disease (SD), partial response (PR), or complete response (CR)) will have both the safety follow-up period and survival follow-up period to occur simultaneously during the 2-year follow-up period. The duration of this follow-up is up to 2 years following the last dose of study treatment, although a longer follow-up period could be considered in selected cases if an efficacy signal is apparent. Patients will receive follow-up CT/MRI scans every 2 months (±14 days) until documented progression of disease, withdrawal of consent from active participation in the study, lost to follow-up, or for at least 2 years after start of treatment, whichever is earliest. Tumor evaluations will be assessed by the investigators and response to be determined according to response evaluation criteria in solid tumors (RECIST) v1.1 guidelines. Tumor assessment scans, for participants who have ongoing clinical benefit beyond the 2-year period from start of treatment, may continue to be collected as part of standard-of-care treatment. Subsequent therapies will also be recorded in this survival follow-up period.

All subjects who discontinue treatment for any reason will have a safety follow-up visit about 30, 60 and 100 days after treatment discontinuation and will be followed for OS and post-study anticancer therapies approximately every 90 days by phone or review of medical records until death, withdrawal of consent, or lost to follow-up.

To minimize the risks of adding or nivolumab + ipilimumab followed by nivolumab and chemo-radiation, safety will be monitored by a Bayesian stopping rule for the rate of treatment-related AEs leading to discontinuation greater than 30% (summarized baseline toxicity rate). For example, if 3 patients out of the first 6 or 4 out of the first 7 evaluable patients experience treatment-related AEs leading to discontinuation, accrual to the trial will be temporarily suspended and the principle investigator and study team will review the toxicity data and recommend either modification or termination of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent

  * Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care
  * Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
* Histological or cytological confirmation of locally advanced or metastatic pancreatic carcinoma prior to entering this study
* No prior chemotherapy regimens received for PC
* Age 18 years or older
* Life expectancy greater than 6 months
* ECOG/WHO Performance Status (PS) 0-1
* All participants will be required to undergo mandatory pre- and on-treatment biopsies at acceptable clinical risk as judged by the investigator. An archival pre-treatment sample is acceptable
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1.5 x 10⁹/L
  * Platelet count ≥ 100 x 10⁹/L
  * Serum bilirubin ≤ 1.5 x upper limit of normal (ULN) (patients with Gilbert's Syndrome must have a total bilirubin ≤ 50 mmol/L)
  * AST/ALT ≤ 5 x ULN
  * Serum creatinine ≤ 1.5 x ULN or CrCl ≥ 40 mL/min (using the Cockcroft-Gault formula)
* Women of child bearing potential (WOCBP) must use method(s) of contraception as indicated in Appendix 3. For a teratogenic study drug and/or when there is insufficient information to assess teratogenicity (preclinical studies have not been done), a highly effective method(s) of contraception (failure rate of less than 1% per year) is required. The individual methods of contraception and duration should be determined in consultation with the investigator. WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 30 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab and ipilimumab is up to 25 days and 18 days, respectively. WOCBP should therefore use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year (Appendix 3). The investigator shall review contraception methods and the time period that contraception must be followed. Men that are sexually active with WOCBP must follow instructions for birth control when the half-life of the investigational drug is greater than 24 hours, contraception should be continued for a period of 90 days plus the time required for the investigational drug to undergo five half-lives. The half-life of nivolumab is up to 25 days. Men who are sexually active with WOCBP must continue contraception for 31 weeks (90 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug. Women who are not of childbearing potential (ie, who are postmenopausal or surgically sterile as well as azoospermic men do not require contraception
* Subjects must have signed and dated a BIOPAC approved written informed consent form in accordance with regulatory and institutional guidelines

Exclusion Criteria:

* Metastatic disease
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results
* Participants with active, known or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participants with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients should be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Allergies and adverse drug reaction

  * History of allergy to study drug components
  * History of severe hypersensitivity reaction to any monoclonal antibody
* WOCBP who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 55 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2024-05-24 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related AEs, SAEs, AEs leading to discontinuation, death, and laboratory abnormalities | 12 months

SECONDARY OUTCOMES:
Median PFS using RECIST v1.1 | 12 months
Median OS | 24 months
Objective Response Rate (ORR) by RECIST v1.1 | 12 months
Rate of downstaging to surgical resection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Inna M Chen, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev & Gentofte University Hospital, Denmark, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No